CLINICAL TRIAL: NCT04160806
Title: The Effect Of Prefrontal Transcranial Direct Current Stimulation On Clinical Severity, Attentional Bias and Interoceptive Accuracy In Panic Disorder
Brief Title: The Effect Of Transcranial Direct Current Stimulation In Panic Disorder
Acronym: PDStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Raşit Tükel, Clinical Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-141
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Panic Disorder
Keywords: Anxiety disorders; Panic disorder; Transcranial Direct Current Stimulation; Interoceptive accuracy; Attention bias; Emotion recognition; Brain Stimulation
MeSH Terms: conditions — Panic Disorder; Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Active Comparator): Left anodal/right anodal transcranial direct current stimulation over the dorsolateral prefrontal cortex
  Interventions: Device: Transcranial direct current stimulation
- Sham Group (Sham Comparator): Sham transcranial direct current stimulation over the dorsolateral prefrontal cortex
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Participants will receive a total of 10 stimulation sessions. During each session, 2 milliAmpers of active or sham tDCS will be applied for 20 minutes over the dorsolateral prefrontal cortex (left anodal/right anodal).
  Other Names: tDCS; Direct current stimulation; transcranial electrical stimulation

SUMMARY:
The aim of the present study is to investigate the effect of prefrontal transcranial Direct Current Stimulation (tDCS) on clinical severity, attentional bias and interoceptive accuracy in panic disorder (PD).

The participants will be assigned to active and sham groups (1:1) and will receive 10 sessions of tDCS. The study will also examine if the effects may last for a month.

DETAILED DESCRIPTION:
Panic Disorder (PD) is one of the most common anxiety disorders. In spite of several available medications, there are unsatisfactory outcomes in a considerable proportion of PD patients and novel treatment approaches are lacking. Given that response to pharmacotherapeutical and psychological treatments occur after long intervals and medications may cause substantial adverse effects which may affect treatment compliance, fast acting and well-tolerated treatments such as non-invasive brain stimulation are considered to be useful as primary treatment approach or as an add-on treatment in PD. Repetitive Transcranial Magnetic Stimulation (rTMS) trials targeting prefrontal cortex mostly reported favorable outcomes in PD.

Transcranial Direct Current Stimulation (tDCS) is another promising non-invasive brain stimulation method with numerous distinctive aspects including its low-cost, robust safety and tolerability, low dropout rates, easy application, reliable blinding procedures and the opportunity to use concomitantly with other treatments. Left anodal/right anodal tDCS over the dorsolateral prefrontal cortex has been demonstrated to decrease attentional bias and amygdala reactivity to threat in individuals with high trait anxiety. Moreover, a treatment-resistant case of PD was reported to have significant amelioration of symptoms up to one month after 10 sessions of tDCS.

The study is a triple-blind randomized controlled trial. The sample will be consisted of thirty participants diagnosed as having PD due to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria. The participants will be assigned to active or sham groups equally. Clinical severity will be assessed with adequate scales. Emotion recognition, attentional bias to threat and interoceptive accuracy will also be measured. Then, participants will be applied ten active or sham sessions of left anodal/right cathodal tDCS over the dorsolateral prefrontal cortex (DLPFC). All measurements will be repeated after the applications. Succinctly, the aim of this study is to assess the effect of ten sessions left anodal/right cathodal tDCS over the DLPFC on clinical severity, attentional bias and interoceptive accuracy in PD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of Panic Disorder, as confirmed by the Structured Clinical Interview for the DSM-5 (SCID-5);
* Patients currently on medication must be at the same stable dose(s) for one month prior to enrollment and be willing to continue at the same dose(s) through the duration of the study;
* Right-hand dominancy assessed by Edinburgh Handedness Inventory;
* Willingness and ability to comply with the requirements of the study protocol;
* Naïve to tDCS.
* 5 or more years of education

Exclusion Criteria:

* Illiteracy, deficient language or refusal to participate or being not able to follow instructions or complete study tasks;
* Less than 5 years of education
* Individuals with any current or lifetime diagnosis of other Axis I disorders, as confirmed by the Structured Clinical Interview for the DSM-5 (SCID-5);
* History of substance or psychoactive compound use,with the exception of nicotine consumption;
* The presence of mental retardation diagnosis (previously identified)
* Individuals with a clinically defined neurological disorder, with an increased risk of seizure for any reason, with a history of treatment with rTMS, deep brain stimulation for any disorder will be excluded;
* Any personal or family history (1st degree relatives) of seizures other than febrile childhood seizures
* Personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes;
* Significant hearing loss or visual impairment;
* Diagnosis of any serious or uncontrolled medical condition such as chronic obstructive pulmonary disease, congestive heart failure or renal failure;
* Skin diseases that could potentially cause irritations under electrodes;
* Patients missing two consecutive protocol sessions;
* Patients with cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Changes in Panic Disorder Severity Scale (PDSS) scores | Up to one month
  The PDSS consists of seven items, each rated on a 5-point scale, which ranges from 0 to 4. The items assess panic frequency, resulting distress, panic-focused anticipatory anxiety, phobic avoidance of situations and of physical sensations, impairment in occupational and social functioning. The overall assessment is made by a total score, which is calculated by summing the scores for all seven items. Minimum score is 0 and maximum score is 28. Higher scores indicate high levels of panic symptomatology. Reduction in score from baseline indicates clinical improvement of panic symptoms.
Changes in Hamilton Anxiety Rating Scale (HAM-A) scores | Up to one month
  The Hamilton Anxiety Rating Scale (HAM-A) is a multiple item questionnaire used to provide an indication of anxiety severity. Higher scores indicate high levels of symptomatology. Minimum score is 0 and maximum score is 56. Reduction in score from baseline indicates clinical symptom improvement.
Changes in Clinical Global Impression-Severity (CGI-S) scores | Up to one month
  Higher scores indicate the presence of high symptom severity. Decrease in scores from baseline reflects clinical symptom improvement. Minimum score is 1 and maximum score is 7. Patients will be classified as responders with a CGI-S = 1 or 2; and partial responders CGI-S = 3.
Changes in performance on an attentional dot-probe task | Up to one month
  Computerized "dot-probe " attentional task will be used. Pairs of emotional faces (neutral/angry or neutral/happy) are randomly presented on a screen. Then, a probe is presented. Subjects are asked to indicate which side the probe approved and need to press the dot after the probe. Total time spent on Region of Interest (angry/neutral face) is measured. Attentional bias towards threat score is the subtraction of median reaction times (milliseconds) in congruent angry versus neutral trials from incongruent angry versus neutral trials. Minimum score is -1000 and maximum score is 1000. Positive scores indicate the presence of attentional vigilance towards threat whereas negative scores indicate an attentional avoidance towards threat.

SECONDARY OUTCOMES:
Changes in Hamilton Depression Rating Scale (HAM-D) scores | Up to one month
  The Hamilton Depression Rating Scale (HAM-D) is a 17-item questionnaire used to provide an indication of depression severity. Minimum score is 0 and maximum score is 52. Higher scores indicate high levels of symptomatology. Reduction in score from baseline indicates clinical symptom improvement.
Changes in Beck Depression Inventory (BDI) scores | Up to one month
  The Beck Depression Inventory is a self-report questionnaire used to provide an indication of depression severity. Minimum score is 0 and maximum score is 63. Higher scores indicate high levels of symptomatology. Reduction in score from baseline indicates clinical symptom improvement.
Changes in Sheehan Disability Scale (SDS) Work/School scores | Up to one month
  The SDS Work/School is a single item measure rated on a 10-point scale. The SDS Work/School measures the extent to which work/school is impaired by symptoms. Minimum score is 0 and maximum score is 10, with higher scores reflecting greater impairment.
Changes in Sheehan Disability Scale (SDS) Social Life scores | Up to one month
  The SDS Social Life is a single item measure rated on a 10-point scale. The SDS Social Life measures the extent to which social life is impaired by symptoms. Minimum score is 0 and maximum score is 10, with higher scores reflecting greater impairment.
Changes in Sheehan Disability Scale (SDS) Family Life/Home Responsibilities scores | Up to one month
  The SDS Family Life/Home Responsibilities is a single item measure rated on a 10-point scale. The SDS Family Life/Home Responsibilities measures the extent to which family life/home responsibilities is impaired by symptoms. Minimum score is 0 and maximum score is 10, with higher scores reflecting greater impairment.
Changes in Body Vigilance Scale (BVS) scores | Up to one month
  BVS is designed to assess conscious attention focused on internal bodily sensations and perturbations. It is an 4-item likert type scale. Minimum score is 0 and maximum score is 40. Higher scores reflect greater body vigilance.
Changes in Heartbeat Detection Accuracy | Up to one month
  Heartbeat detection accuracy is an index ranging between 0 and 1 showing heart rate prediction performance. Higher scores reflect better interoceptive abilities. Heartbeat detection (interoceptive) accuracy is calculated by the following equation: 1/N ∑ (1 - (|recorded heartbeats - counted heartbeats|)/recorded heartbeats). N was the number of blocks for the heartbeat detection task.
Changes in the number of correct responses at a facial expression recognition task | Up to one month
  Participants are presented with individual pictures of facial expressions of emotions. Each presented face displays one of six basic emotions (anger, disgust, fear, happiness, sadness, or surprise). Each emotional expression is presented at different levels of intensity which have been created by combining shape and texture features of the two extremes "neutral" (0%) and "full prototypical emotion" (100%) to varying degrees. Participants are instructed to correctly classify each facial expression as angry, disgusted, fearful, happy, sad, surprised or neutral. Responses are made by pushing one out of six labelled keys on a response box. Hit rates and false alarm rates are measured separately for each emotion. Minimum accuracy percentage of an emotion is 0 and maximum accuracy percentage of an emotion is 100. Higher accuracy rates indicate better emotion recognition.

CONTACTS AND LOCATIONS:
Overall Officials: Raşit Tükel, Professor, Principal Investigator — Istanbul University
Locations (1):
- Department Of Psychiatry, Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No